CLINICAL TRIAL: NCT02970019
Title: A Double-blind, Placebo-controlled Study to Determine Safety, Tolerability, Pharmacokinetic of K0706.
Brief Title: Safety and Tolerability Study of K0706 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_16_27
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- K0706 (Experimental): K0706 will be administered once a day
  Interventions: Drug: K0706
- Placebo (Experimental): Placebo will be administered once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K0706 — Once a day administration after fast
  Arms: K0706
Drug: Placebo — Once a day administration after fast
  Arms: Placebo

SUMMARY:
This is a safety, tolerability and pharmacokinetic study in subjects with Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written, and dated, informed consent (or legally acceptable representative/impartial witness when applicable) and is available for the entire study
2. Willing and able to comply with the scheduled visits, treatment plan, laboratory testing, study procedures, and restrictions (in the Investigator's opinion), and be accessible for follow-up
3. Male or female aged 18 to 65 years (both inclusive)
4. Diagnosed with Parkinson's disease

Exclusion Criteria:

1. Clinical diagnosis of genetic form of Parkinson's disease, or drug-induced parkinsonism
2. Diagnosis of Parkinson's disease Dementia (probable, possible)
3. Presence of severe dyskinesias
4. History of brain surgery for Parkinson's disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Adverse events | 4 weeks

SECONDARY OUTCOMES:
Peak plasma concentration | 4 weeks
Area under the plasma concentration versus time curve | 4 weeks
Time of observed peak plasma concentration | 4 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - SPARC Site 03, Long Beach, California
  - SPARC Site 05, Panorama City, California
  - SPARC Site 01, DeLand, Florida
  - SPARC Site 02, Orlando, Florida
  - SPARC Site 04, Raleigh, North Carolina

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102